CLINICAL TRIAL: NCT01180335
Title: Randomized Trial Comparing Standard Neoadjuvant Chemotherapy to Genomic Driven Chemotherapy Regimen in Patients With Breast Cancer
Brief Title: Standard Neoadjuvant Chemotherapy Versus Genomic Driven Chemotherapy in Patients With Breast Cancer
Acronym: REMAGUS04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Institut Curie (Other)
Responsible Party: ANDRE Fabrice, G.I.E. REMAGUS
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CSET1376
Record Dates: First submitted 2010-08-05; First posted 2010-08-12 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2010-08

CONDITIONS: Breast Cancer
Keywords: Genomic driven chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Active Comparator): 4 cycles FEC followed by 4 cycles docetaxel
  Interventions: Drug: Chemotherapy
- Genomic driven chemotherapy (Experimental): High DLD30 receive 3 months weekly paclitaxel followed by 4 FEC, patients with high TOP2A receive 4FEC then 4 docetaxel, patients with low DLD30 and low TOP2A are treated with 6 cycles of docetaxel-capecitabine.
  Interventions: Drug: Genomic driven chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — 4 cycles FEC followed by 4 cycles docetaxel
  Arms: Chemotherapy
Drug: Genomic driven chemotherapy — High DLD30 receive 3 months weekly paclitaxel followed by 4 FEC, patients with high TOP2A receive 4FEC then 4 docetaxel, patients with low DLD30 and low TOP2A are treated with 6 cycles of docetaxel-capecitabine.
  Arms: Genomic driven chemotherapy

SUMMARY:
This randomized trial is comparing a standard neoadjuvant chemotherapy with a genomic driven chemotherapy in patients with breast cancer.

DETAILED DESCRIPTION:
After a core biopsy, each tumor is profiled using Affymetrix U133plus2 gene expression array. DLD30 score (Hess, JCO, 2006) and TOP2A expression are quantified. Patients are then either treated with 4FEC followed by 4 docetaxel (standard arm) or by a genomic-driven regimen (experiemental arm). In the experimental arm, patients with high DLD30 receive 3 months weekly paclitaxel followed by 4 FEC, patients with high TOP2A receive 4FEC then 4 docetaxel, patients with low DLD30 and low TOP2A are treated with 6 cycles of docetaxel-capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer not eligible for conservative surgery
* Her2 negative
* Amount of tumor cells >30% on HES slides
* RIN>6 and amount of RNA>1 ug
* No metastases
* Subject, age > 18 years and <65 years old
* Signed written informed consent
* PS 0-1
* No previous treatment for breast cancer
* Adequate organ function
* FEVG >50%

Exclusion Criteria:

* In situ carcinoma
* Multifocal cancers
* Her2+
* Presence of metastasis
* Genomic testing not feasible because of tumor cells <30%, RIN<6, insufficient amount of RNA
* Organ dysfunction that contraindicates chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Complete response rate based on the histology | Tumoral assessment at 4 and 8 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Florence LEREBOURS, MD, Principal Investigator — Centre René Huguenin; Jean-Yves PIERGA, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Gustave Roussy, Villejuif, France